CLINICAL TRIAL: NCT00124748
Title: A Randomized Open-label Study of 400 mg Versus 800 mg of Imatinib Mesylate in Patients With Newly Diagnosed, Previously Untreated Chronic Myeloid Leukemia in Chronic Phase (CML-CP) Using Molecular Endpoints.
Brief Title: Efficacy of 400 Mg Versus 800 Mg Imatinib in Chronic Myeloid Leukemia in Chronic Phase Patients - TOPS (Tyrosine Kinase Inhibitor Optimization and Selectivity)
Acronym: TOPS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was prematurely discontinued because no improvement was observed in the 800mg dose compared to 400mg dose
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571K2301; NCT00324636 (obsolete NCT alias)
Record Dates: First submitted 2005-07-27; First posted 2005-07-28 (Estimated); Results first posted 2012-02-03 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-01

CONDITIONS: Leukemia, Myeloid, Chronic Phase
Keywords: CML; Philadelphia positive; Bcr-abl; imatinib mesylate; Chronic myeloid leukemia (CML) in chronic phase
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

ARMS (2):
- Imatinib 400 mg (Experimental): Oral dose of 400mg Imatinib once daily. All patients received the assigned dose starting on Day 0 (Visit 3). The dose of Imatinib could be interrupted, reduced, or escalated based on guidelines defined in protocol.
  Interventions: Drug: Imatinib mesylate
- imatinib 800 mg (Experimental): Patients randomized to receive 800 mg Imatinib were to receive 400 mg twice daily (b.i.d.) oral administration, in the morning and the evening. All patients received the assigned dose starting on Day 0 (Visit 3). The dose of Imatinib could be interrupted or reduced based on guidelines defined in protocol.
  Interventions: Drug: Imatinib mesylate

INTERVENTIONS:
Drug: Imatinib mesylate — Imatinib is packaged in bottles as 100mg and 400mg tablets
  Other Names: STI571; Gleevec; Glivec

SUMMARY:
This study investigated the safety and efficacy of 400mg Versus 800mg imatinib in patients with newly diagnosed, previously untreated chronic myeloid leukemia in chronic phase (CML-CP) using molecular endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Patients within 6 months of diagnosis (date of initial diagnosis is the date of first cytogenetic analysis)
* Diagnosis of chronic myelogenous leukemia (CML) in chronic phase with cytogenetic confirmation of Philadelphia chromosome of (9;22) translocations and presence of Breakpoint cluster region gene-abelson proto-oncogene (Bcr-Abl)
* Documented chronic phase CML
* Adequate end organ function as defined by:

  * total bilirubin < 1.5 x Upper Limit of Normal (ULN)
  * Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) < 2.5 x ULN
  * creatinine < 1.5 x ULN

Exclusion Criteria:

* Patients in late chronic phase, accelerated phase, or blastic phase are excluded
* Patients who have received other investigational agents
* Patients who received Gleevec/Glivec for any duration prior to study entry, with the exception of those patients successfully completing [CSTI571A2107 (NCT00428909)] study immediately prior to the participation in this study
* Patient received any treatment for CML prior to study entry for longer than 2 weeks with the exception of hydroxyurea and/or anagrelide
* Patients with another primary malignancy except if the other primary malignancy is neither currently clinically significant or requiring active intervention
* Patients who are: (a) pregnant, (b) breast feeding, (c) of childbearing potential without a negative pregnancy test prior to baseline and (d) male or female of childbearing potential unwilling to use barrier contraceptive precautions throughout the trial (post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential).
* Patient with a severe or uncontrolled medical condition (i.e., uncontrolled diabetes,chronic renal disease)
* Patient previously received radiotherapy to ≥ 25% of the bone marrow
* Patient had major surgery within 4 weeks prior to study entry, or who have not recovered from prior major surgery
* Patients with an Eastern Cooperative Oncology Group (ECOG) Performance Status Score ≥ 3
* Patients with International normalized ratio (INR) or partial thromboplastin time (PTT) > 1.5 x ULN, with the exception of patients on treatment with oral anticoagulants
* Patients with known positivity for human immunodeficiency virus (HIV); baseline testing for HIV is not required
* Patients with identified sibling donors where allogeneic bone marrow transplant is elected as first line treatment

Other protocol-defined inclusion/exclusion criteria applied.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2005-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (74):
- United States (49):
  - University of South Alabama, Mobile, Alabama
  - Alta Bates Comprehsenive Cancer Center, Berkeley, California
  - University of Miami, Berkeley, California
  - South Bay Oncology Hematology Partners, Campbell, California
  - UCLA Medical Center, Los Angeles, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Osler Medical Inc., Melbourne, Florida
  - Advanced Medical Specialists, Miami, Florida
  - Integrated Community Oncology Network, Orange Park, Florida
  - Hematology-Oncology Associates, P.A., Pensacola, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - Indiana Blood and Marrow Institutw, Beech Grove, Indiana
  - Indiana Blood and Marrow Transplant, Beech Grove, Indiana
  - University of Iowa Hospitals & Clinic, Iowa City, Iowa
  - University of Kentucky - C201 Clinic, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Lousville Oncology, Clinical Research Program M-25, Louisville, Kentucky
  - Jayne S. Gurtler, MD, Laura A. Brinz, MD & Angelo Russo, MD, Metairie, Louisiana
  - Hematology and Oncology Specialists, New Orleans, Louisiana
  - LSU Health Science Center, Shreveport, Louisiana
  - LSU Health Scine Center, Shreveport, Louisiana
  - St. Agnes Hospital, Baltimore, Maryland
  - Great Lakes Cancer Institute, Lansing, Michigan
  - U of Minnesota, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cancer Center of the Carolinas, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University Hospitals of Cleveland, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Kaiser Permanente Northwest Region Oncology/Hemacology, Portland, Oregon
  - Kaiser Permanente Northwest Region, Portland, Oregon
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburg, Hillman Cancer Center, Pittsburgh, Pennsylvania
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - Cancer Center of the Carolinas, Greenville, South Carolina
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - The Jones Clinic, Germantown, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - UT Southwestern Harold C. Simmons Comprehensive Cancer Center, Dallas, Texas
  - University of Texas / MD Anderson Cancer Center, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Virgina Cancer Center, UVA Division of Hematology & Oncology, Charlottesville, Virginia
- Argentina (2):
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, La Plata
- Australia (12):
  - Novartis Investigative Site, St Leonards, New South Wales
  - Novartis Investigative Site, Waratah, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, East Melbourne, Victoria
  - Novartis Investigative Site, Fitzroy, Victoria
  - Novartis Investigative Site, Frankston, Victoria
  - Novartis Investigative Site, Parkville, Victoria
  - Novartis Investigative Site, Prahran, Victoria
  - Novartis Investigative Site, South Brisbane
- Novartis Investigative Site, Campinas, Brazil
- Canada (4):
  - Novartis Investigative Site, Calgary
  - Novartis Investigative Site, Montreal
  - Novartis Investigative Site, Ottawa
  - Novartis Investigative Site, Québec
- Italy (6):
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Florence
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Orbassano
  - Novartis Investigative Site, Roma

REFERENCES:
- [Derived] Branford S, Yeung DT, Parker WT, Roberts ND, Purins L, Braley JA, Altamura HK, Yeoman AL, Georgievski J, Jamison BA, Phillis S, Donaldson Z, Leong M, Fletcher L, Seymour JF, Grigg AP, Ross DM, Hughes TP. Prognosis for patients with CML and >10% BCR-ABL1 after 3 months of imatinib depends on the rate of BCR-ABL1 decline. Blood. 2014 Jul 24;124(4):511-8. doi: 10.1182/blood-2014-03-566323. Epub 2014 May 23. PMID 24859364
- [Derived] Branford S, Yeung DT, Ross DM, Prime JA, Field CR, Altamura HK, Yeoman AL, Georgievski J, Jamison BA, Phillis S, Sullivan B, Briggs NE, Hertzberg M, Seymour JF, Reynolds J, Hughes TP. Early molecular response and female sex strongly predict stable undetectable BCR-ABL1, the criteria for imatinib discontinuation in patients with CML. Blood. 2013 May 9;121(19):3818-24. doi: 10.1182/blood-2012-10-462291. Epub 2013 Mar 20. PMID 23515925
- [Derived] Guilhot F, Hughes TP, Cortes J, Druker BJ, Baccarani M, Gathmann I, Hayes M, Granvil C, Wang Y. Plasma exposure of imatinib and its correlation with clinical response in the Tyrosine Kinase Inhibitor Optimization and Selectivity Trial. Haematologica. 2012 May;97(5):731-8. doi: 10.3324/haematol.2011.045666. Epub 2012 Feb 7. PMID 22315495
- See also: Visit NovartisClinicalTrials.com: Pre-qualify for a trial, and view a list of trials and participating study centers. — http://www.novartisclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Imatinib 400 mg: Oral dose of 400mg Imatinib once daily (q.d.). All patients received the assigned dose starting on Day 0 (Visit 3). The dose of Imatinib could be interrupted, reduced, or escalated based on guidelines defined in protocol.
Period: Overall Study
Arm/Group | Imatinib 400 mg | Imatinib 800 mg
Started | 157 | 319
Safety Population | 157 | 316
Completed | 14 | 35
Not Completed | 143 | 284
Not completed — Adverse Event | 8 | 39
Not completed — Abnormal laboratory Value | 2 | 2
Not completed — Abnormal Procedure | 0 | 1
Not completed — Lack of Efficacy | 20 | 41
Not completed — No longer requires study drug | 1 | 1
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 5 | 15
Not completed — Lost to Follow-up | 2 | 7
Not completed — Administrative Problem(Study Terminated) | 101 | 174
Not completed — Death | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Imatinib 400 mg | Imatinib 800 mg | Total
Number analyzed (Participants) | 157 | 319 | 476
Age Continuous [Mean (Standard Deviation); unit: years] | 46.2 (14.90) | 48.2 (13.89) | 47.6 (14.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 136 | 209
  Male | 84 | 183 | 267

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Major Molecular Response (MMR) Rates at 12 Months
Description: MMR is defined as Bcr-Abl (A fusion gene of the breakpoint cluster region [Bcr] gene and Abelson proto-oncogene [Abl] genes) transcript ratio ≤0.1% (≥ 3 log reduction of BCR-ABL transcripts from a standardized baseline), as detected by reverse transcriptase polymerase chain reaction [RT-PCR] (performed centrally).
Time Frame: 12 months
Population: Intent-to-treat (ITT) population consisted of all patients who are randomized into the study.
Measure: Number; unit: Percentage of participants
Arm/Group | Imatinib 400 mg | Imatinib 800 mg
Number analyzed (Participants) | 157 | 319
Percentage of participants | 38.9 | 45.1

2. Secondary Outcome: Percentage of Participants With Major Molecular Response (MMR) Rates at 24, 36, and 42 Months
Description: as for outcome 1
Time Frame: 24, 36 and 42 months
Population: Intent-to-treat (ITT) population consisted of all patients who are randomized into the study.
Measure: Number; unit: Percentage of participants
Arm/Group | Imatinib 400 mg | Imatinib 800 mg
Number analyzed (Participants) | 157 | 319
Percentage of participants
  24 months | 53.5 | 50.8
  36 months | 52.2 | 49.8
  42 months | 51.6 | 50.2

3. Secondary Outcome: Percentage of Participants With Complete Cytogenetic Response (CCyR) Rate at 12, 24, 36, 42 Months
Description: Cytogenetic response (CyR)is the percentage of Philadelphia chromosome positive metaphases (among at least 20 metaphase cells in bone marrow (BM)) with Complete Cytogenetic Response (CCyR) being 0 percent.
Time Frame: 12, 24, 36, 42 months
Population: Intent-to-treat (ITT) population consisted of all patients who are randomized into the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | Imatinib 400 mg | Imatinib 800 mg
Number analyzed (Participants) | 157 | 319
Percentage of Participants
  12 months | 66.9 | 70.2
  24 months | 76.4 | 76.8
  36 months | 79.0 | 80.6
  42 months | 80.3 | 81.5

4. Secondary Outcome: Percentage of Participants With Complete Hematological Response (CHR) Rates at 12, 24, 36, and 42 Months
Description: Complete Hematologic Response (CHR) is where all of the following criteria must be present for ≥4 weeks: White Blood Cell (WBC) count <10 x 109/L, Platelet count <450 x 109/L, Basophils <5%, No blasts and promyelocytes in Peripheral Blood (PB), (Myelocytes + metamyelocytes) < 5% in PB and No evidence of extramedullary involvement.
Time Frame: 12, 24, 36, and 42 months
Population: Intent-to-treat (ITT) population consisted of all patients who are randomized into the study.
Measure: Number; unit: Percentage of participants
Arm/Group | Imatinib 400 mg | Imatinib 800 mg
Number analyzed (Participants) | 157 | 319
Percentage of participants
  12 months | 94.9 | 93.7
  24 months | 94.9 | 93.7
  36 months | 96.2 | 94.4
  42 months | 96.2 | 94.4

5. Secondary Outcome: Percentage of Patients With Undetectable Levels of Bcr-Abl (A Fusion Gene of the Breakpoint Cluster Region [Bcr] Gene and Abelson Proto-oncogene [Abl] Genes) Transcripts
Description: "Undetectable levels" or Complete molecular response is defined as Bcr-Abl ratio (%) on international scale (IS) <= 0.0032% (≥ 4.5 log reduction of BCR-Abl transcripts from a standardized baseline).
Time Frame: 12 , 24, 36 and 42 months
Population: Intent-to-treat (ITT) population consisted of all patients who were randomized into the study.
Measure: Number; unit: Percentage of Partcipants
Arm/Group | Imatinib 400 mg | Imatinib 800 mg
Number analyzed (Participants) | 157 | 319
Percentage of Partcipants
  12 Months | 4.5 | 4.7
  24 Months | 11.5 | 10.3
  36 Months | 12.7 | 13.2
  42 Months | 14.6 | 12.5

6. Secondary Outcome: Time to First Major Molecular Response
Description: MMR is defined as Bcr-Abl (A fusion gene of the breakpoint cluster region [Bcr] gene and Abelson proto-oncogene [Abl] genes) transcript ratio ≤0.1% (≥ 3 log reduction of BCR-ABL transcripts from a standardized baseline), as detected by reverse transcriptase polymerase chain reaction [RT-PCR] (performed centrally).
  Time to MMR (months) = (date of first MMR or censoring - date of randomization + 1) / 30.4375. Time to first MMR was evaluated using the Kaplan-Meier method
Time Frame: 42 months overall
Population: Intent-to-treat (ITT) population consisted of all patients who were randomized to the study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib 400 mg | Imatinib 800 mg
Number analyzed (Participants) | 157 | 319
Months | 13.6 [10.8 to 15.6] | 8.4 [8.3 to 9.0]

7. Secondary Outcome: Time to First Complete Cytogenetic Response
Description: Cytogenetic response (CyR) is the percentage of Philadelphia positive metaphases (among at least 20 metaphase cells in Bone Marrow) with Complete Cytogenetic Response (CCyR) being 0 percent. Time to CCyR (months) = (date of first CCyR or censoring - date of randomization + 1) / 30.4375. Time to first CCyR was evaluated using the Kaplan-Meier method.
Time Frame: 60 months overall
Population: Intent-to-treat (ITT) population consisted of all patients who are randomized into the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib 400 mg | Imatinib 800 mg
Number analyzed (Participants) | 157 | 319
Months | 10.8 [5.9 to 11.2] | 5.8 [5.8 to 6.0]

8. Secondary Outcome: Time to First Complete Hematological Response (CHR)]
Description: Complete Hematological Response (CHR) is defined is where all of the following criteria must be present for ≥4 weeks: White Blood Cell (WBC) count <10 x 109/L, Platelet count <450 x 109/L, Basophils <5%, No blasts and promyelocytes in Peripheral Blood (PB), (Myelocytes + metamyelocytes) < 5% in PB and No evidence of extramedullary involvement. Time to CHR (months) = (date of first CHR or censoring - date of randomization + 1) / 30.4375. Time to first CHR was evaluated using the Kaplan-Meier method.
Time Frame: 60 months overall
Population: Intent-to-treat (ITT) population consisted of all patients who are randomized into the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib 400 mg | Imatinib 800 mg
Number analyzed (Participants) | 157 | 319
Months | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]

9. Secondary Outcome: Estimated Rate of Event Free Survival (EFS) in Two Treatment Arms
Description: EFS on treatment was defined as time between randomization and either (1) death due to any cause during study treatment, (2) progression to accelerated phase (AP) or blast crisis (BC) on treatment, (3) loss of complete hematological response (CHR), or (4) loss of major cytogenic response (MCyR) while on treatment. Estimated rate of EFS was analyzed by Kaplan-Meier estimate (percent probability and 95% Confidence interval).
Time Frame: 60 months over all
Population: Intent-to-treat (ITT) population consisted of all patients who are randomized into the study.
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Imatinib 400 mg | Imatinib 800 mg
Number analyzed (Participants) | 157 | 319
Percent probability
  12 Months | 95.3 [90.5 to 97.7] | 98.0 [95.6 to 99.1]
  24 Months | 94.6 [89.5 to 97.3] | 95.3 [92.1 to 97.3]
  36 Months | 92.3 [86.5 to 95.7] | 94.5 [91.1 to 96.7]
  42 Months | 92.3 [86.5 to 95.7] | 94.1 [90.5 to 96.3]
  48 Months | 92.3 [86.5 to 95.7] | 93.6 [89.9 to 96.0]
  60 Months | 90.3 [82.7 to 94.7] | 93.6 [89.9 to 96.0]

10. Secondary Outcome: Estimated Rate of Progression Free Survival (PFS) in Two Treatment Arms
Description: PFS on study which was defined as time between randomization and either (1) death due to any cause on treatment of during follow-up after discontinuation of treatment or (2) progression to accelerated phase (AP) or blast crisis (BC) on treatment during follow-up after discontinuation of study treatment. Estimated rate of PFS was analyzed by Kaplan-Meier estimate (percent probability and 95% Confidence interval).
Time Frame: 60 months over all and follow up period
Population: Intent-to-treat (ITT) population consisted of all patients who are randomized into the study.
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Imatinib 400 mg | Imatinib 800 mg
Number analyzed (Participants) | 157 | 319
Percent probability
  12 Months | 97.4 [93.2 to 99.0] | 98.7 [96.5 to 99.5]
  24 Months | 95.9 [91.2 to 98.2] | 97.5 [94.9 to 98.8]
  36 Months | 94.4 [89.0 to 97.1] | 96.7 [93.7 to 98.3]
  42 Months | 94.4 [89.0 to 97.1] | 96.3 [93.2 to 98.0]
  48 Months | 94.4 [89.0 to 97.1] | 95.8 [92.5 to 97.7]
  60 Months | 94.4 [89.0 to 97.1] | 95.8 [92.5 to 97.7]

11. Secondary Outcome: Estimated Rate of Progression to Accelerated Phase (AC)/Blast Crisis (BC) in Two Treatment Arms
Description: (Accelerated Phase/Blast Crisis) AP/BC was defined as time between randomization and either (1) (Chronic Myeloid Leukemia) CML-related death (if death was primary reason for discontinuation) or (2) progression to AP or BC (during treatment). Estimated rate of AC/BC was analyzed by Kaplan-Meier estimate (percent probability and 95% Confidence interval).
Time Frame: 60 months over all and follow up period
Population: Intent-to-treat (ITT) population consisted of all patients who are randomized into the study.
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Imatinib 400 mg | Imatinib 800 mg
Number analyzed (Participants) | 157 | 319
Percent probability
  12 Months | 97.4 [93.2 to 99.0] | 99.0 [97.0 to 99.7]
  24 Months | 95.9 [91.2 to 98.2] | 97.9 [95.3 to 99.0]
  36 Months | 95.2 [90.1 to 97.7] | 97.5 [94.7 to 98.8]
  42 Months | 95.2 [90.1 to 97.7] | 97.0 [94.1 to 98.5]
  48 Months | 95.2 [90.1 to 97.7] | 97.0 [94.1 to 98.5]
  60 Months | 95.2 [90.1 to 97.7] | 97.0 [94.1 to 98.5]

12. Secondary Outcome: Estimated Rate of Overall Survival (OS) in Two Treatment Arms
Description: OS was defined as time between randomization and death due to any cause during study treatment or during follow-up after discontinuation of treatment. Estimated rate of OS was analyzed by Kaplan-Meier estimate (percent probability and 95% Confidence interval).
Time Frame: 60 months over all and follow up period
Population: Intent-to-treat (ITT) population consisted of all patients who are randomized into the study.
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Imatinib 400 mg | Imatinib 800 mg
Number analyzed (Participants) | 157 | 319
Percent probability
  12 Months | 98.7 [94.9 to 99.7] | 99.0 [97.1 to 99.7]
  24 Months | 97.4 [93.2 to 99.0] | 97.8 [95.4 to 98.9]
  36 Months | 96.1 [91.4 to 98.2] | 95.5 [92.5 to 97.3]
  42 Months | 94.7 [89.7 to 97.2] | 94.8 [91.6 to 96.8]
  48 Months | 94.0 [88.7 to 96.8] | 93.4 [89.7 to 95.8]
  60 Months | 94.0 [88.7 to 96.8] | 93.4 [89.7 to 95.8]

13. Secondary Outcome: Kaplan-Meier Estimates of Duration of First Major Molecular Response Until Confirmed Loss
Description: Duration of MMR (months) = (date of first confirmed loss or censoring - date of MMR + 1 ) / 30.4375. Estimated rate of duration of first MMR was analyzed by Kaplan-Meier estimate (percent probability and 95% Confidence interval).
Time Frame: From First major molecular response to first confirmed loss or censoring
Population: Intent-to-treat (ITT) population consisted of all patients who are randomized into the study.
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Imatinib 400 mg | Imatinib 800 mg
Number analyzed (Participants) | 157 | 319
Percent probability
  3 Months | 100 [100 to 100] | 96.3 [92.9 to 98.0]
  6 Months | 98.3 [93.3 to 99.6] | 90.7 [86.2 to 93.8]
  9 Months | 97.4 [92.2 to 99.2] | 90.2 [85.7 to 93.4]
  12 Months | 95.6 [89.8 to 98.2] | 88.4 [83.6 to 91.9]
  15 Months | 93.8 [87.4 to 97.0] | 87.5 [82.5 to 91.2]
  18 Months | 92.8 [86.2 to 96.4] | 86.1 [80.9 to 90.0]
  21 Months | 90.9 [83.8 to 95.0] | 85.1 [79.8 to 89.1]
  24 Months | 89.9 [82.5 to 94.3] | 83.6 [78.0 to 87.8]
  30 Months | 88.5 [80.5 to 93.4] | 82.5 [76.8 to 86.9]
  36 Months | 85.1 [75.6 to 91.1] | 81.1 [75.1 to 85.8]
  42 Months | 85.1 [75.6 to 91.1] | 77.9 [70.4 to 83.8]

14. Secondary Outcome: Kaplan-Meier Estimates of Duration of First Complete Cytogenetic Response (CCyR)
Description: Duration of CCyR was defined as the time between date of CCyR and the earliest of either (1) loss of CCyR OR (2) (Chronic Myeloid Leukemia) CML-related death or progression to (Accelerated Phase/Blast Crisis) AP/BC during study treatment. Estimated rate of duration of first CCyR was analyzed by Kaplan-Meier estimate (percent probability and 95% Confidence interval).
Time Frame: From first complete cytogenetic response to first confirmed loss or censoring
Population: Intent-to-treat (ITT) population consisted of all patients who are randomized into the study.
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Imatinib 400 mg | Imatinib 800 mg
Number analyzed (Participants) | 157 | 319
Percent probability
  6 Months | 99.1 [94.0 to 99.9] | 99.2 [96.7 to 99.8]
  12 Months | 98.2 [93.1 to 99.6] | 97.8 [94.7 to 99.1]
  18 Months | 98.2 [93.1 to 99.6] | 97.3 [94.1 to 98.8]
  24 Months | 98.2 [93.1 to 99.6] | 96.8 [93.3 to 98.4]
  30 Months | 98.2 [93.1 to 99.6] | 96.8 [93.3 to 98.4]
  36 Months | 98.2 [93.1 to 99.6] | 95.9 [91.9 to 98.0]
  42 Months | 98.2 [93.1 to 99.6] | 95.9 [91.9 to 98.0]

15. Secondary Outcome: Mean Actual Dose Intensity Per Day
Description: The mean actual dose intensity per day from start of treatment up to last dose or discontinuation was evaluated up to Month 36. Actual dose intensity (mg/day) = total dose/time on treatment (periods of zero dose are included)
Time Frame: start of treatment to Month 36
Population: Safety analysis population (SAP): consisted of all patients who received at least one dose of study medication.Subjects are summarized according to the safety treatment allocation (the dose they actually received).
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Imatinib 400 mg | Imatinib 800 mg
Number analyzed (Participants) | 157 | 316
mg/day | 399.3 (83.84) | 643.3 (158.63)

16. Secondary Outcome: Imatinib Pharmacokinetic Trough Plasma Concentration (Cmin) at Month 12
Description: Imatinib PK trough plasma concentration (Cmin) was defined as any pre-dose Imatinib plasma concentration
Time Frame: Month 12
Population: Pharmakokinetic (PK) population consisted of number of patients with a pre-dose PK sample at Month 12
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Imatinib 400 mg | Imatinib 800 mg
Number analyzed (Participants) | 86 | 150
mg/mL | 1458.2 (2259.5) | 739.58 (1321.09)

17. Secondary Outcome: Estimated Rates of Progression Free Survival (PFS) on Treatment by Major Molecular Response (MMR)
Description: A Landmark Kaplan-Meier analysis was performed for PFS at 42 months by MMR status at 6, 12, and 18 months to investigate their prognostic value.
Time Frame: 42 months
Population: Intent-to-treat (ITT) population consisted of all patients who were randomized to the study treatment. Patients without a valid polymerase chain reaction (PCR) assessment or those who had experienced an event before the landmark were excluded from analysis
Measure: Number (95% Confidence Interval); unit: Percent probability
Arm/Group | Imatinib 400 mg | Imatinib 800 mg
Number analyzed (Participants) | 134 | 274
Percent probability
  No MMR at 6 Months | 94.8 [88.0 to 97.8] | 95.6 [90.3 to 98.0]
  MMR at 6 Months | 100 [100 to 100] | 99.0 [93.2 to 99.9]
  No MMR at 12 Months | 93.2 [82.9 to 97.4] | 94.6 [87.4 to 97.7]
  MMR at 12 Months | 100 [100 to 100] | 99.3 [95.0 to 99.9]
  No MMR at 18 Months | 96.7 [78.6 to 99.5] | 97.0 [88.6 to 99.3]
  MMR at 18 Months | 98.7 [91.2 to 99.8] | 99.3 [95.2 to 99.9]

18. Secondary Outcome: Time to First Complete Molecular Response (CMR)]
Description: Complete Molecular Response is defined as a Bcr-Abl (a fusion of gene of Bcr and ABl genes) ratio ≤0.0032% on the International Scale Bcr = breakpoint cluster gene Abl = abelson proto-oncogene.
Time Frame: 48 months overall
Population: This analysis was not done because no major molecular improvement was observed in the 800mg dose compared to 400mg dose. Hence, analysis for complete molecular response was not necessary.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Imatinib 400 mg | Imatinib 800 mg
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Number of Participants With the Effect of Imatinib on the Diabetic Participants With Known Concomitant Type II Diabetes
Time Frame: 12 months
Population: Due to the small number of diabetic patients enrolled into the study, the analysis was never done.
Measure: Number; unit: Participants
Arm/Group | Imatinib 400 mg | Imatinib 800 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Imatinib 400mg: Oral dose of 400mg imatinib once daily. All patients received the assigned dose starting on Day 0 (Visit 3). The dose of Imatinib could be interrupted, reduced, or escalated based on guidelines defined in protocol.
- Imatinib 800mg: Patients randomized to receive 800 mg imatinib were to receive 400 mg twice daily (b.i.d.) oral administration, in the morning and the evening. All patients received the assigned dose starting on Day 0 (Visit 3). The dose of Imatinib could be interrupted or reduced based on guidelines defined in protocol.
Arm/Group | Imatinib 400mg | Imatinib 800mg
Serious Adverse Events (participants affected / at risk) | 42/157 | 121/316
Other Adverse Events (participants affected / at risk) | 157/157 | 315/316
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib 400mg (N=157) | Imatinib 800mg (N=316)
Anaemia (Blood and lymphatic system disorders) | 3 | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 5
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 5 | 12
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Splenic cyst (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 9
Angina pectoris (Cardiac disorders) | 2 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 3
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac discomfort (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 0 | 1
Phimosis (Congenital, familial and genetic disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1
Amaurosis (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 0 | 2
Retinal detachment (Eye disorders) | 0 | 2
Retinal haemorrhage (Eye disorders) | 0 | 1
Retinal vein occlusion (Eye disorders) | 0 | 1
Uveitis (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Anal polyp (Gastrointestinal disorders) | 0 | 1
Caecitis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 4
Diverticulum (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 2
Gastritis alcoholic (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3
Haematemesis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 2
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 3
Reflux gastritis (Gastrointestinal disorders) | 0 | 1
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 4
Adverse drug reaction (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 2
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 2 | 0
Concomitant disease progression (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Device ineffective (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Polyp (General disorders) | 0 | 1
Polyserositis (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 13
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 2
Hepatotoxicity (Hepatobiliary disorders) | 0 | 2
Liver disorder (Hepatobiliary disorders) | 1 | 1
Appendicitis (Infections and infestations) | 0 | 5
Bacterial infection (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 3
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 5
Gastroenteritis viral (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1
HIV infection (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 5
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Retroperitoneal abscess (Infections and infestations) | 0 | 1
Salmonellosis (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 1 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 2
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Electrocardiogram T wave abnormal (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Blast crisis in myelogenous leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Desmoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Cervical myelopathy (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
IIIrd nerve paralysis (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 1 | 1
Nerve root compression (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 3
Parkinsonism (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 3
Transient ischaemic attack (Nervous system disorders) | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 1 | 0
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Neonatal disorder (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Placental disorder (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Premature labour (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 2
Calculus ureteric (Renal and urinary disorders) | 0 | 3
Calculus urinary (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Paroxysmal nocturnal haemoglobinuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Urethral disorder (Renal and urinary disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 4
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Pregnancy of partner (Social circumstances) | 2 | 2
Circulatory collapse (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib 400mg (N=157) | Imatinib 800mg (N=316)
Anaemia (Blood and lymphatic system disorders) | 41 | 120
Leukopenia (Blood and lymphatic system disorders) | 20 | 51
Neutropenia (Blood and lymphatic system disorders) | 38 | 107
Thrombocytopenia (Blood and lymphatic system disorders) | 36 | 111
Conjunctival haemorrhage (Eye disorders) | 8 | 19
Conjunctivitis (Eye disorders) | 9 | 19
Eye swelling (Eye disorders) | 3 | 19
Eyelid oedema (Eye disorders) | 21 | 45
Lacrimation increased (Eye disorders) | 8 | 30
Periorbital oedema (Eye disorders) | 46 | 132
Abdominal discomfort (Gastrointestinal disorders) | 13 | 17
Abdominal distension (Gastrointestinal disorders) | 9 | 15
Abdominal pain (Gastrointestinal disorders) | 36 | 76
Abdominal pain upper (Gastrointestinal disorders) | 38 | 54
Constipation (Gastrointestinal disorders) | 19 | 36
Diarrhoea (Gastrointestinal disorders) | 71 | 184
Dyspepsia (Gastrointestinal disorders) | 21 | 57
Flatulence (Gastrointestinal disorders) | 7 | 20
Gastritis (Gastrointestinal disorders) | 6 | 20
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 28
Haemorrhoids (Gastrointestinal disorders) | 6 | 25
Nausea (Gastrointestinal disorders) | 78 | 205
Toothache (Gastrointestinal disorders) | 14 | 21
Vomiting (Gastrointestinal disorders) | 54 | 140
Asthenia (General disorders) | 22 | 48
Chest pain (General disorders) | 9 | 7
Chills (General disorders) | 9 | 18
Face oedema (General disorders) | 13 | 64
Fatigue (General disorders) | 51 | 131
Influenza like illness (General disorders) | 12 | 35
Oedema (General disorders) | 10 | 35
Oedema peripheral (General disorders) | 43 | 135
Pyrexia (General disorders) | 31 | 75
Bronchitis (Infections and infestations) | 10 | 26
Gastroenteritis (Infections and infestations) | 8 | 26
Influenza (Infections and infestations) | 17 | 18
Nasopharyngitis (Infections and infestations) | 19 | 30
Pharyngitis (Infections and infestations) | 5 | 17
Sinusitis (Infections and infestations) | 13 | 33
Upper respiratory tract infection (Infections and infestations) | 44 | 88
Urinary tract infection (Infections and infestations) | 17 | 26
Contusion (Injury, poisoning and procedural complications) | 6 | 18
Procedural pain (Injury, poisoning and procedural complications) | 7 | 16
Alanine aminotransferase increased (Investigations) | 11 | 25
Aspartate aminotransferase increased (Investigations) | 11 | 26
Platelet count decreased (Investigations) | 1 | 18
Weight decreased (Investigations) | 6 | 26
Weight increased (Investigations) | 26 | 54
Decreased appetite (Metabolism and nutrition disorders) | 22 | 54
Fluid retention (Metabolism and nutrition disorders) | 3 | 21
Hypocalcaemia (Metabolism and nutrition disorders) | 8 | 28
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 33
Hypophosphataemia (Metabolism and nutrition disorders) | 30 | 43
Arthralgia (Musculoskeletal and connective tissue disorders) | 48 | 107
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 71
Bone pain (Musculoskeletal and connective tissue disorders) | 17 | 39
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 16
Muscle spasms (Musculoskeletal and connective tissue disorders) | 69 | 141
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 10 | 14
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 22 | 29
Myalgia (Musculoskeletal and connective tissue disorders) | 37 | 83
Neck pain (Musculoskeletal and connective tissue disorders) | 10 | 16
Pain in extremity (Musculoskeletal and connective tissue disorders) | 33 | 79
Dizziness (Nervous system disorders) | 38 | 47
Dysgeusia (Nervous system disorders) | 8 | 37
Headache (Nervous system disorders) | 46 | 98
Paraesthesia (Nervous system disorders) | 11 | 16
Anxiety (Psychiatric disorders) | 12 | 24
Depression (Psychiatric disorders) | 20 | 32
Insomnia (Psychiatric disorders) | 21 | 53
Cough (Respiratory, thoracic and mediastinal disorders) | 34 | 74
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 44
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 21
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 27
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 38
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 18
Night sweats (Skin and subcutaneous tissue disorders) | 18 | 25
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 41
Rash (Skin and subcutaneous tissue disorders) | 32 | 119
Hypertension (Vascular disorders) | 12 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.